CLINICAL TRIAL: NCT06817889
Title: An Open-Label Study to Assess the Safety and Efficacy of Remdesivir for Treatment of Symptomatic Laboratory-Confirmed Respiratory Syncytial Virus Infection of the Upper Respiratory Tract in Patients Receiving Cellular or Bispecific Antibody Therapies
Brief Title: Remdesivir for the Treatment of Upper Respiratory Tract Infection Due to RSV in Immunocompromised Individuals
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125015; NCI-2025-00572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20650 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Autoimmune Disease; Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Autoimmune Diseases; Respiratory Syncytial Virus Infections | interventions — remdesivir; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (remdesivir) (Experimental): Patients receive remdesivir IV over 30-120 minutes on days 1-5, with the option to extend to day 10 at the investigator's discretion, in the absence of disease progression or unacceptable toxicity. Patients also undergo nasal swabs and blood sample collection throughout the study.
  Interventions: Drug: Remdesivir; Other: Survey Administration; Procedure: Biospecimen Collection; Procedure: Nasal Swab

INTERVENTIONS:
Drug: Remdesivir — Given IV
  Other Names: 2-Ethylbutyl (2S)-2-(((S)-(((2R,3S,4R,5R)-5-(4-aminopyrrolo(2,1-f)(1,2,4)triazin-7-yl)-5-cyano-3,4-dihydroxytetrahydrofuran-2-yl)methoxy)(phenoxy)phosphoryl)amino)propanoate; GS-5734; L-Alanine, N-((S)-hydroxyphenoxyphosphinyl)-, 2-Ethylbutyl Ester, 6-Ester with 2-C-(4-aminopyrrolo(2,1-f)(1,2,4)triazin-7-yl)-2,5-anhydro-D-altrononitrile; RDV; SARS-CoV-2 antiviral agents: remdesivir; Veklury
Other: Survey Administration — Ancillary studies
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Nasal Swab — Undergo nasal swabs
  Other Names: Nasal Swab Test; Nasopharyngeal Swab; Nasopharyngeal Swab Test

SUMMARY:
This phase II trial tests how well remdesivir works for treatment of respiratory syncytial virus (RSV) infection of the upper respiratory tract in patients receiving cellular or bispecific antibody therapy. Cellular or bispecific antibody therapies cause suppression of the immune system, making infections more frequent and reducing the body's ability to fight the infections. RSV infections are one of the most common respiratory infections in immunocompromised individuals and can cause significant pneumonia and even death. Remdesivir is in a class of medications called antivirals. It works by stopping viruses from spreading in the body.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive remdesivir intravenously (IV) over 30-120 minutes on days 1-5, with the option to extend to day 10 at the investigator's discretion, in the absence of disease progression or unacceptable toxicity. Patients also undergo nasal swabs and blood sample collection throughout the study.

After completion of study treatment, patients are followed up on day 14 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent (where locally approved)
* RSV confirmed by local lab testing via nucleic acid amplification test (e.g. polymerase chain reaction [PCR] or respiratory viral panel [RVP]) using an upper respiratory tract sample collected within the 5 days prior to day 1 (RDV dosing)
* Symptomatic RSV infection of the upper respiratory tract, with symptom onset and positive microbiologic testing within the 5 days prior to day 1 (RDV dosing). Symptomatic RSV infection is defined as having new upper respiratory symptom(s) or worsening of a pre-existing upper respiratory symptom (if chronic and associated with a previously existing diagnosis, such as chronic lung disease, chronic rhinorrhea, or seasonal allergies)
* Have a hematologic malignancy and/or autoimmune disease and received one of the following treatments relative to RSV diagnosis date:

  * Received allogeneic hematopoietic cell transplant (HCT) with any conditioning regimen within 1 year
  * Received autologous HCT with any conditioning regimen within 3 months
  * Received Chimeric antigen receptor T cell therapy (CARTx) within 3 months
  * Received bispecific antibody therapy (bsAb) within 3 months
* Categorized as moderate-risk (overall score 3-6) or high-risk (overall score 7-10) per an adapted version of the Immunodeficiency Scoring Index (ISI) for RSV, as below, relative to the day of RSV diagnosis:

  * 1 point:

    * Recent (within the prior 30 days) allogeneic HCT, autologous HCT, or CARTx
    * Corticosteroids within the prior 30 days for management of graft versus host disease (GVHD) or cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS).
  * 2 points:

    * Age ≥ 40 years
  * 3 points:

    * Absolute neutrophil count (ANC) < 500 cells/μL within the prior 7 days
    * Absolute lymphocyte count (ALC) < 200 cells/µL within the prior 7 days
* Oxygen saturation (SpO2) 93% or greater on room air and at rest (to be measured after participant has rested in a quiet room for ≥ 2 minutes, with oxygen [O2] saturation probe on finger or earlobe for ≥ 1 minute, with saturation reading remaining ≥ 93%) at screening
* Willingness to take study drug and complete necessary study procedures
* Participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception as described

Exclusion Criteria:

* Received or receiving an approved or authorized direct-acting antiviral therapy with potential efficacy against RSV (e.g. ribavirin) for ≥ 24 hours within the prior 7 days, and/or expected to receive anti-RSV direct-acting antiviral therapies for RSV during the course of the study at the time of screening
* Received or receiving investigational direct-acting antiviral therapies against RSV for the current RSV episode
* Received any investigational anti-RSV monoclonal antibodies or off-label use of approved anti-RSV monoclonal antibodies within < 4 months or < 5 half-lives, whichever is longer, before screening, or expected to receive anti-RSV monoclonal antibodies during the course of the study at the time of screening
* Received an RSV vaccine after cellular therapy or after starting the current antitumor therapeutic regimen
* Participation in any other concurrent clinical trial of an experimental treatment for RSV, including RSV vaccines
* Alanine aminotransferase (ALT) ≥ 5 times the upper limit of normal within 7 days prior to screening
* New lower respiratory tract radiographic abnormalities or clinical symptoms after RSV-associated symptom onset that are suspected to be due to RSV
* Unable to tolerate nasal sampling required for this study, as determined by the investigator (e.g., history of significant epistaxis, nasopharyngeal anatomical abnormalities, nasal or sinus surgery)
* A life expectancy of three months or less, as determined by the investigator
* Pregnant, as determined by a Point-of-Care urine pregnancy test or reported by the patient or their electronic health record within 7 days of screening
* Receiving, requiring, or expected to require supplemental oxygen for RSV-related illness or SpO2 < 93% at rest < 24 hours prior to study drug administration
* Previous infection and/or hospitalization for RSV, or previous infection with, treatment for, or hospitalization for another respiratory viral infection within 28 days prior to screening
* Documented positive test for other respiratory viruses concomitantly (limited to influenza, parainfluenza, adenovirus, human metapneumovirus, or coronavirus [including SARS-CoV-2]) ≤ 7 days prior to screening, as determined by local testing (additional testing not required)
* Clinically significant bacteremia or fungemia ≤ 7 days prior to screening and not adequately treated, as determined by the investigator
* Clinically significant bacterial, fungal, or viral pneumonia within two (2) weeks prior to screening and not adequately treated, as determined by the investigator
* Clinically significant symptoms of CRS or ICANS within the prior 72 hours before screening that is not adequately controlled, as determined by the investigator
* Any inability to take study drug or comply with study procedures that, in the opinion of the investigator, would make the participant unsuitable for the study
* Known hypersensitivity or allergy to the study drug, its metabolites, or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants requiring ≥ 2 liters/minute of oxygen for ≥ 24 consecutive hours | Up to day 29
  Will be estimated with 95% Wilson confidence intervals.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) and laboratory abnormalities | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Incidence of serious adverse events and AEs leading to study drug discontinuation | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Proportion of participants with RSV-related hospitalization (if not hospitalized at the time of first dose) or death | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Supplemental oxygen free days | Up to day 29
  Defined as days alive and not requiring ≥ 2 liters/minute of supplemental oxygen. Will be compared between cohorts using weighted least squares linear regression with propensity score weights.
Proportion of participants who develop new or worsening pulmonary infiltrates | Up to day 29
  Based on radiographic imaging of the lungs for standard of care.
Proportion of participants requiring high-flow nasal cannula, non-invasive ventilation, or invasive mechanical ventilation for ≥ 24 consecutive hours | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Proportion of participants admitted to intensive care unit | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Proportion of participants who die | Up to day 29
  Will consider using time-to-event methods such as cumulative incidence curves and Cox proportional hazards regression.
Change from baseline in RSV nasal swab viral load | From baseline through day 3 and 5
  Will be computed among participants with baseline nasal viral loads ≥ the lower limit of quantitation and compared between cohorts using linear regression with propensity score weights.
Maximum daily Respiratory Infection Intensity and Impact Questionnaire (RiiQ) score | From baseline to day 29
  The RiiQ is a 13-item questionnaire, with each item representing a different RSV-associated symptom and graded on a 4-point scale (0 = None, 1 = Mild, 2 = Moderate, and 3 = Severe). Greater scores indicate greater symptom severity. Recall period is the past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hill, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No